CLINICAL TRIAL: NCT07078422
Title: Home Use Study of Targeted Mechanical Stimulation for Tremor Relief
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Encora, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20232333
Record Dates: First submitted 2025-04-09; First posted 2025-07-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Essential Tremor; Parkinson's Disease
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: The study design is modeled after a typical movement assessment, relevant to the diagnosis, and modified to apply the treatment. Participants will perform movements typical of the motor assessments both before and during treatment. The intent of the study is to confirm the device design and usability in the subject's home environment. The study will also measure change in treatment effect after long periods of regular use.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- A (Experimental): Oder of assessment begins with TETRAS and ends with ADLs
  Interventions: Device: Encora Pulse
- B (Experimental): Order of assessment begins with ADLs and ends with TETRAs
  Interventions: Device: Encora Pulse
- C (Experimental): Order of assessment begins with TETRAS and ends with ADLs, but both are administered backwards
  Interventions: Device: Encora Pulse
- D (Experimental): Order of assessment begins with ADLs and ends with TETRAs, but both are administered backwards
  Interventions: Device: Encora Pulse

INTERVENTIONS:
Device: Encora Pulse — The proposed therapeutic device is a wristband that delivers personalized therapeutic relief to users by adjusting parameters of mechanical vibration, tailored to each individual user's tremor. It measures and characterizes users' upper limb tremor before determining what parameters of mechanical vibration should be applied to stimulate the sensory neurons on the wrist.
  This study will not be conducted under IDE. It is a non-significant risk due to the non-invasive nature of mechanical vibration.

SUMMARY:
Subjects will receive prototype devices to be used for participation. The study comprises three phases:

1. Alpha phase: Two remote study visits and an in-home period to gather device usability data on the alpha system. The at home period for this phase will be 2 weeks. This phase will be used to confirm that the device and labeling are suitable for in-home use.
2. Beta Phase B1: Beta Phase B1 will be conducted using the beta devices for two in-person or remote, 60 to 90-minute, visits. This phase will be used to assess design changes between alpha and beta versions.
3. Beta Phase B2: Seven remote visits and in-home usage to gather usability and efficacy data on the beta system in-home. Beta Phase B2 will be conducted using the beta devices for 12 weeks. This phase will be used to assess design changes between alpha and beta versions.

ELIGIBILITY:
Inclusion Criteria - Alpha and Beta Phase B1

* Age 18 years or older, able to comply with all study procedures and capable of providing informed consent.
* Mentally competent to understand and able to perform written, informed consent to participate in the study
* A diagnosis of either ET or PD as determined by clinical history
* Moderate to severe upper limb tremor

Exclusion Criteria - Alpha and Beta Phase B1

* Pregnant women
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
* History of psoriasis, eczema or atopic dermatitis at the stimulation site
* History of peripheral neuropathy in the upper limbs, including carpal tunnel syndrome and diabetic neuropathy
* Participant unable to communicate with sponsor/investigator and staff
* Any other medical conditions or physical or mental impairments that in the sponsor/investigator's opinion would render the subject unsuitable as a candidate for the study.

Inclusion Criteria - Beta Phase B2

* Age 18 years or older, able to comply with all study procedures and capable of providing informed consent
* Mentally competent to understand and able to perform written, informed consent to participate in the study
* For ET subjects, a diagnosis of essential tremor defined as definite or probable ET based on TRIG criteria
* For PD subjects, a diagnosis of Parkinson's disease by a Movement Disorder Specialist
* For ET subjects, at least one hand exhibiting tremor > 2 as assessed by the Essential Tremor Rating Assessment Scale (TETRAS) finger to nose task, duck wing task, OR Archimedes Spiral completed during the Screening visit
* For PD subjects, a score > 2 on at least one of MDS-UPDRS items 3.15, 3.16 or 3.17 At the Screening Visit, a score of > 3 on one of the following subject-assessed items of the Bain & Findley Activities of Daily Living Scale (BF-ADL): Use a spoon to drink soup, Hold a cup of tea, Do up buttons, Do up a zipper, Write a letter
* Stable medications for at least 30 days prior to enrollment and the ability to maintain tremor medications throughout the duration of study participation
* For PD subjects, able to participate in visits in a practically defined OFF state (withdrawal from all tremor medication for 12 hours prior to study visits)
* A wrist circumference of 6.0 - 8.1 inches

Exclusion Criteria - Beta Phase B2

* Pregnant women
* Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site
* History of psoriasis, eczema or atopic dermatitis at the stimulation site
* History of peripheral neuropathy in the upper limbs, including carpal tunnel syndrome and -diabetic neuropathy
* Participant unable to communicate with sponsor/investigator and staff
* Any other medical conditions or physical or mental impairments that in the sponsor/investigator's opinion would render the subject unsuitable as a candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Assess the design changes between the alpha and beta versions of the device | Data will be collected at baseline and visit one.
  This outcome measure assesses participants' experiences through an open-ended survey. Participants will be asked to describe their perceptions, symptoms, and overall experiences with the treatment. No predefined responses are given, and answers will be analyzed qualitatively
To assess the usability of the beta device in an at-home setting | Data will be collected at baseline, week 1, week 2, month 1, month 2 and month 3.
  Characterization of any unforeseen errors during subject interaction with the packaging device and instructions for use during at-home use will be collected using the usability survey which is an open ended, qualitative survey that measures patient usage error and device related satisfaction

SECONDARY OUTCOMES:
To establish the quantitative efficacy in upper limb tremor reduction using the BF-ADL scale | Data will be collected at baseline, week 1, week 2, month 1, month 2 and month 3.
  The Bain and Findley Tremor ADL Scale (BF-ADL) is a tool used to assess the impact of essential tremor on a person's ability to perform activities of daily living (ADLs), specifically those involving the upper limbs. The effectiveness of the device in reducing limb tremor will be evaluated using the BF-ADL scale. The scale rates each activity on a 1-to-4 scale: 1 indicates the activity can be done without difficulty, 2 with little effort, 3 with a lot of effort, and 4 means the activity cannot be done alone.
To establish the quantitative efficacy in upper limb tremor reduction using the TETRAS scale | Data will be collected at baseline, week 1, week 2, month 1, month 2 and month 3.
  The effectiveness of the device in reducing limb tremor will be evaluated using the TETRAS (Tremor Research Group Essential Tremor Rating Assessment Scale) tool. Tremor severity will be measured on a scale of 0 to 4; a score of 0 indicates no tremor, while a score of 4 represents severe tremor. Scores between 0 and 4 can be assigned using increments of 0.5, allowing for a more nuanced assessment of tremor severity.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Murray, MD, Principal Investigator — WVU Comprehensive Movement Disorder Clinic
Locations (1):
- Encora Therapeutics, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No